CLINICAL TRIAL: NCT02764905
Title: A Comprehensive Intervention for Promoting Successful Aging Amongst Below the Cognitive Norm Older People With Diabetes- a Feasibility Study
Brief Title: Intensive Cognitive and Physical Rehabilitation Program
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Tali Cukierman-Yaffe, M.D, Sheba Medical Center
Other Study IDs: SHEBA-16-2953-TCY-CTIL
Record Dates: First submitted 2016-05-01; First posted 2016-05-06 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Cognitive Rehabilitation; Physical Rehabilitation
Keywords: Diabetes; Cognitive-physical rehabilitation; Self care management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intensive cognitive-physical rehabilitation group: will include a 2 phase multi-disciplinary intervention. The 2 phases: a) Intensive phase: weekly 4 hour group meeting which will include computerized cognitive training, aerobic, balance and strength exercise and group discussion that will be dedicated to cognitive rehabilitation strategies development and implementation with emphasis on disease management and physical activity as well as psycho-education on various disease management aspects (medical and nutritional) b) a consolidation phase: monthly 2 hour group discussions on challenges of implementation and coping strategies
  Interventions: Behavioral: intensive cognitive physical rehabilitation program

INTERVENTIONS:
Behavioral: intensive cognitive physical rehabilitation program — include 2 phases: a) Intensive phase: weekly 4 hour group meeting which will include computerized cognitive training, aerobic, balance and strength exercise and group discussion that will be dedicated to cognitive rehabilitation strategies development and implementation with emphasis on disease management and physical activity as well as psycho-education on various disease management aspects (medical and nutritional) b) a consolidation phase: monthly 2 hour group discussions on challenges of implementation and coping strategies.

SUMMARY:
This will be a feasibility study. Individuals that have undergone an evaluation day at the center for successful aging with diabetes with a Glycosylated hemoglobin (A1C) of >=7.5 and a Montreal Cognitive Assessment (MoCA)<26 will be approached and invited to participate. The participants will be divided into 2 groups: 1) information communication technology (ICT) group - an intervention based on weekly SMS that will remind the individual to implement his personal treatment plan and will raise the awareness to the importance of self-care in diabetes; 2) intensive cognitive-physical rehabilitation group that will include a 2 phase multi-disciplinary intervention. The 2 phases: a) Intensive phase: weekly 4 hour group meeting which will include computerized cognitive training, aerobic, balance and strength exercise and group discussion that will be dedicated to cognitive rehabilitation strategies development and implementation with emphasis on disease management and physical activity as well as psycho-education on various disease management aspects (medical and nutritional) b) a consolidation phase: monthly 2 hour group discussions on challenges of implementation and coping strategies. Outcomes will include change in A1C (primary), change in strength, aerobic capacity as well as quality of life and cognitive function (secondary). Additionally, team members and participants will fill out a structured questionnaire regarding their evaluation of the program aiming at refinement of the intervention.

DETAILED DESCRIPTION:
Intensive cognitive-physical rehabilitation intervention. The intervention will include two phases:

1. Intensive phase: 12 weekly group meeting 4 hours each. Each meeting will be composed of:

   * 2 hours guided by a neuropsychologist each dedicated to a different cognitive domain for example memory, concentration, planning, information processing, problem solving (with special emphasis on diabetes issues). Each session will be composed of: 1) introduction- homework from previous session will be checked and the cognitive domain that will be discussed on that day will be introduced; 2) cognitive training using a computerized system (hour); 3) group discussion on compensatory strategies and training to be conducted at home
   * 2 hours guided by a certified physical trainer. These will include strength, balance and aerobic elements conducted in a group but individualized according to the capabilities and targets of the individual as assessed during the evaluation day. These sessions will also include formulation of a plan for exercise to be conducted by the individual on a daily basis. Additionally, 30 minutes of each session will be dedicated to psycho-education on various disease management aspects guided by a diabetes nurse educator or a dietitian (alternating).
2. Consolidation phase: 9 months of monthly group meetings. The consolidation group sessions will include monthly 2 hour group discussions on challenges of implementation and coping strategies Medical surveillance will take place every 2 months with monitoring of glucose, blood pressure lipid control as well as follow-up on other recommendations given during the feed-back sessions this will be conducted by the Diabetes nurse educator who will be work together with a diabetes specialist an Endocrinologist (study physician) on maximal risk factor reduction.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diabetes above the age of 65 and
* with a MoCA score of below 26
* with a A1C>=7.5% .
* All the individuals will be Hebrew speaking without significant hearing or visual disability.

Exclusion Criteria:

* Diagnosed dementia or cognitive impairment
* Any major non-diabetes related illness expected to reduce life expectancy substantially or interfere with study participation and illiterate individuals to participate in the study.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with type 2 diabetes with below the norm cognitive function
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
change in A1C | 3 months, 12 months
  obtained from the results of routine lab tests conducted in the individual's respective health maintenance organization (HMO)

SECONDARY OUTCOMES:
change in indices will be collected before initiation of intervention and will be measured again after 3 months and 12 months | 3 months, 12 months
  The 6 min walk test score
change in indices will be collected before initiation of intervention and will be measured again after 3 months and 12 months | 3 months, 12 months
  Grip strength using a Jammer dynamometer
change in indices will be collected before initiation of intervention and will be measured again after 3 months and 12 months | 3 months, 12 months
  Change in quality of life (WHO-5 wellbeing questionnaire, the single general self- rated health question)

CONTACTS AND LOCATIONS:
Overall Officials: Tali Cukierman-yaffe, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cukierman T, Gerstein HC, Williamson JD. Cognitive decline and dementia in diabetes--systematic overview of prospective observational studies. Diabetologia. 2005 Dec;48(12):2460-9. doi: 10.1007/s00125-005-0023-4. Epub 2005 Nov 8. PMID 16283246
- [Background] Biessels GJ, Deary IJ, Ryan CM. Cognition and diabetes: a lifespan perspective. Lancet Neurol. 2008 Feb;7(2):184-90. doi: 10.1016/S1474-4422(08)70021-8. PMID 18207116
- [Background] Reijmer YD, van den Berg E, Ruis C, Kappelle LJ, Biessels GJ. Cognitive dysfunction in patients with type 2 diabetes. Diabetes Metab Res Rev. 2010 Oct;26(7):507-19. doi: 10.1002/dmrr.1112. PMID 20799243
- [Background] Exalto LG, Biessels GJ, Karter AJ, Huang ES, Katon WJ, Minkoff JR, Whitmer RA. Risk score for prediction of 10 year dementia risk in individuals with type 2 diabetes: a cohort study. Lancet Diabetes Endocrinol. 2013 Nov;1(3):183-90. doi: 10.1016/S2213-8587(13)70048-2. Epub 2013 Aug 20. PMID 24622366
- [Background] Volpato S, Leveille SG, Blaum C, Fried LP, Guralnik JM. Risk factors for falls in older disabled women with diabetes: the women's health and aging study. J Gerontol A Biol Sci Med Sci. 2005 Dec;60(12):1539-45. doi: 10.1093/gerona/60.12.1539. PMID 16424285
- [Background] Kirkman MS, Briscoe VJ, Clark N, Florez H, Haas LB, Halter JB, Huang ES, Korytkowski MT, Munshi MN, Odegard PS, Pratley RE, Swift CS. Diabetes in older adults. Diabetes Care. 2012 Dec;35(12):2650-64. doi: 10.2337/dc12-1801. Epub 2012 Oct 25. No abstract available. PMID 23100048
- [Background] Punthakee Z, Miller ME, Launer LJ, Williamson JD, Lazar RM, Cukierman-Yaffee T, Seaquist ER, Ismail-Beigi F, Sullivan MD, Lovato LC, Bergenstal RM, Gerstein HC; ACCORD Group of Investigators; ACCORD-MIND Investigators. Poor cognitive function and risk of severe hypoglycemia in type 2 diabetes: post hoc epidemiologic analysis of the ACCORD trial. Diabetes Care. 2012 Apr;35(4):787-93. doi: 10.2337/dc11-1855. Epub 2012 Feb 28. PMID 22374637
- [Background] Sinclair AJ, Girling AJ, Bayer AJ. Cognitive dysfunction in older subjects with diabetes mellitus: impact on diabetes self-management and use of care services. All Wales Research into Elderly (AWARE) Study. Diabetes Res Clin Pract. 2000 Dec;50(3):203-12. doi: 10.1016/s0168-8227(00)00195-9. PMID 11106835
- [Background] Anderson RM, Funnell MM, Butler PM, Arnold MS, Fitzgerald JT, Feste CC. Patient empowerment. Results of a randomized controlled trial. Diabetes Care. 1995 Jul;18(7):943-9. doi: 10.2337/diacare.18.7.943. PMID 7555554
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Stellefson M, Dipnarine K, Stopka C. The chronic care model and diabetes management in US primary care settings: a systematic review. Prev Chronic Dis. 2013;10:E26. doi: 10.5888/pcd10.120180. PMID 23428085
- [Background] Liang X, Wang Q, Yang X, Cao J, Chen J, Mo X, Huang J, Wang L, Gu D. Effect of mobile phone intervention for diabetes on glycaemic control: a meta-analysis. Diabet Med. 2011 Apr;28(4):455-63. doi: 10.1111/j.1464-5491.2010.03180.x. PMID 21392066
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Ropponen A, Silventoinen K, Tynelius P, Rasmussen F. Association between hand grip/body weight ratio and disability pension due to musculoskeletal disorders: a population-based cohort study of 1 million Swedish men. Scand J Public Health. 2011 Dec;39(8):830-8. doi: 10.1177/1403494811424610. Epub 2011 Oct 3. PMID 21969330
- [Background] Yoshida H, Nishi M, Watanabe N, Fujiwara Y, Fukaya T, Ogawa K, Kim MJ, Lee S, Shinkai S. [Predictors of frailty development in a general population of older adults in Japan using the Frailty Index for Japanese elderly patients]. Nihon Ronen Igakkai Zasshi. 2012;49(4):442-8. doi: 10.3143/geriatrics.49.442. Japanese. PMID 23269023
- [Background] Hajos TR, Pouwer F, Skovlund SE, Den Oudsten BL, Geelhoed-Duijvestijn PH, Tack CJ, Snoek FJ. Psychometric and screening properties of the WHO-5 well-being index in adult outpatients with Type 1 or Type 2 diabetes mellitus. Diabet Med. 2013 Feb;30(2):e63-9. doi: 10.1111/dme.12040. PMID 23072401
- [Background] DeSalvo KB, Bloser N, Reynolds K, He J, Muntner P. Mortality prediction with a single general self-rated health question. A meta-analysis. J Gen Intern Med. 2006 Mar;21(3):267-75. doi: 10.1111/j.1525-1497.2005.00291.x. Epub 2005 Dec 7. PMID 16336622
- [Background] Hochberg I, Feraru G, Kozdoba M, Mannor S, Tennenholtz M, Yom-Tov E. Encouraging Physical Activity in Patients With Diabetes Through Automatic Personalized Feedback via Reinforcement Learning Improves Glycemic Control. Diabetes Care. 2016 Apr;39(4):e59-60. doi: 10.2337/dc15-2340. Epub 2016 Jan 28. No abstract available. PMID 26822328